CLINICAL TRIAL: NCT01257633
Title: Observational Study on Surgical Treatment of Early Stage (T1-T2) Glotto-supraglottic Laryngeal Cancer Via Transoral Resection With Robotic Assistance
Brief Title: Surgical Treatment of Early Stage Glotto-supraglottic Laryngeal Cancer Via Transoral Resection With Robotic Assistance
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: AOI/2010/BL-01; 2010-A01190-39 (Other: ANSM)
Record Dates: First submitted 2010-12-09; First posted 2010-12-10 (Estimated); Last update posted 2025-11-17 (Actual); Status verified 2015-03

CONDITIONS: Laryngeal Neoplasms
Keywords: da Vinci surgical robot; laryngeal cancer
MeSH Terms: conditions — Laryngeal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- The study population: Laryngeal cancer patients requiring surgical tumor resection.
  Interventions: Procedure: Transoral robot-assisted tumor resection using the da Vinci robot

INTERVENTIONS:
Procedure: Transoral robot-assisted tumor resection using the da Vinci robot — Transoral robot-assisted tumor resection using the da Vinci robot

SUMMARY:
The main objective of this study is to determine the rate of healthy surgical margins after tumor resection in transoral robot-assisted surgery for glottic and/or supraglottic early stage (T1-T2) laryngeal cancer.

ELIGIBILITY:
Inclusion Criteria:

* The subject has signed consent
* The subject must be a member or beneficiary of a health insurance plan
* The patient is available for 12 months of follow-up
* The subject has a cancer of the larynx:
* classified T1 or T2 in the TNM
* glottic localization and / or supraglottic regardless of node status
* with or without a history of head and neck cancer
* The subject does not have distant metastasis (M0)
* A decision for endoscopic robot-assisted surgery is retained in multidisciplinary meeting

Exclusion Criteria:

-

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is aimed at all patients with early stage (T1 or T2) glottic and / or supraglottic squamous cell carcinoma of the larynx, whatever their status and cervical lymph nodes without distant metastases (M0) and for whom endoscopic surgical treatment with robotic assistance is indicated following a multidisciplinary meeting.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2011-04; Primary Completion 2014-09-30 (Actual); Study Completion 2014-09-30 (Actual)

PRIMARY OUTCOMES:
The presence/absence of cancerous tissue in the surgical margins of the resectioned tumors | 1 day

SECONDARY OUTCOMES:
Time to prepare the surgical setting (min) | 1 day
Time necessary to dock the robot (min) | 1 day
Total surgical time (console time) (min) | 1 day
Intervention time taking into account cervical ganglions (min) | 1 day
Was a tracheotomy necessary? yes/no | 1 day
Presence / absence of bleeding complications | 1 day
Was a conversion to an open procedure necessary? yes/no | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Lallemant, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (3):
- France (3):
  - CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, Gard
  - CHU de Montpellier - Hôpital Gui de Chauliac, Montpellier
  - CHRU de Toulouse - Hôpital de Rangueil, Toulouse

REFERENCES:
- [Result] Lallemant B, Moriniere S, Ceruse P, Lebalch M, Aubry K, Hans S, Dolivet G, Malard O, Bonduelle Q, Vergez S. Transoral robotic surgery for squamous cell carcinomas of the posterior pharyngeal wall. Eur Arch Otorhinolaryngol. 2017 Dec;274(12):4211-4216. doi: 10.1007/s00405-017-4771-9. Epub 2017 Oct 14. PMID 29032418